CLINICAL TRIAL: NCT05393323
Title: Effects of Cervical Distraction Versus Cervical Traction Techniques on Pain, Range of Motion and Function in Patients With Upper Cervical Pain
Brief Title: Effects of Cervical Distraction Versus Cervical Traction Techniques on Upper Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/0136 Hafsa Khan
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: Cervical pain; Traction; Distraction
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distraction technique (Experimental): conventional physical therapy with distraction technique
  Interventions: Other: conventional physical therapy with distraction technique
- Traction technique (Experimental): conventional physical therapy with traction technique
  Interventions: Other: conventional physical therapy with traction technique

INTERVENTIONS:
Other: conventional physical therapy with distraction technique — Distraction will be at suboccipital level and patients will ask to assume a supine position with the head on the plinth. The therapist will use fingertips in both hands from digits 2 through 5, and cups the suboccipital region of the patient and supports the posterior skull. The therapist provides a light distraction to the posterior skull. Distraction will be applied for 10 min with pull for 10 sec and5 sec will be applied. Prior to apply this technique all patients will receive 15 minutes of infrared with TENS at cervical spine. The total treatment session will be of 25 minute with total intervention period of 4 weeks with 5 sessions per week.
  Arms: Distraction technique
Other: conventional physical therapy with traction technique — In cervical traction, patients will ask to lie supine on the treatment table. Head will cradle by physiotherapist from chin and the occiput, and then the physiotherapist will apply traction force in 25 degree neck flexion. Traction will be applied for 10 minutes with pull for 10 sec and 5 sec rest will be applied. Prior to apply this technique all patients will receive 15 minutes of infrared with TENS at cervical spine. The total treatment session will be of 25 min with total intervention period of 4 weeks with 5 sessions per week. All outcome measurements will be assessed before treatment and then reassessed at the end of 4th week.
  Arms: Traction technique

SUMMARY:
The aim of this study is to compare the effects of cervical distraction versus cervical traction techniques on pain, range of motion and function in patients with upper cervical pain. This study will be randomized clinical trial and 42 patients according to inclusion criteria will be included in the study. They will be allocated into 2 groups by non-probability purposive sampling technique. Group A will receive cervical distraction technique with conventional physical therapy while Group B will receive cervical traction technique with conventional therapy. Outcome measures; Neck Disability Index, goniometry and Numeric Pain Rating Scale will measure neck function and neck pain intensity. Both groups will receive 5 sessions per week for 4 weeks and measurements will be taken at the baseline and at the end of 4th week. Data will be analyzed by SPSS version 25

DETAILED DESCRIPTION:
The term collectively used for musculoskeletal conditions originating from cervical area is known as neck pain. According to the Global burden of disease (2010) study, neck pain is the fourth agent which is the reason behind chronic disability. The incidence of cervical pain in the adult population aged 15 to 74 years is 5.92% to 38.7% and it is more prevalent in women than men. The best predictor of future neck pain is the presence of an episode of neck pain in the past. Cervical rotation deficits are noted mostly in upper cervical spine issues as in atlantoaxial joint pathology.

The aim of this study is to compare the effects of cervical distraction versus cervical traction techniques on pain, range of motion and function in patients with upper cervical pain. This study will be a randomized clinical trial and 42 patients according to inclusion criteria will be included in the study. They will be allocated into 2 groups by non-probability purposive sampling technique. Group A will receive the cervical distraction technique with conventional physical therapy while Group B will receive the cervical traction technique with conventional therapy. Outcome measures; Neck Disability Index, goniometry and Numeric Pain Rating Scale will measure neck function and neck pain intensity. Both groups will receive 5 sessions per week for 4 weeks and measurements will be taken at the baseline and at the end of 4th week. Data will be analyzed by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 3 months chronicity of upper cervical pain
* Positive ﬂexion-rotation test (asymmetry of >10◦ between sides or less than 32◦ in any direction)
* hypomobility in one or more segments of C0-1, C1-2, or C2-3

Exclusion Criteria:

* Congenital abnormalities (Cervical torticollis)
* Past surgical history of cervical spine
* Any history of neck trauma
* Already undergone physiotherapy treatment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain
NDI | 4th Week
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50.
Goniometric measurement | 4th Week
  The science of measuring the joint ranges in each plane of the joint is called goniometry. Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. Neck flexion, extension, side bending and rotation will be assessed through it

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Mehmooda begum medical complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaishy S, Kondal S. Effect of Vertical Cervical traction Combined with Conventional Neurodynamic Mobilization and SNAGs in an Individual with Neck Pain and Cervical Radiculopathy: A Case Report.
- [Background] Khan K, Yasmeen S, Ishaque F, Imdad F, Shaikh SA, Nawaz U, et al. A RANDOMIZED CONTROLLED TRIAL TO INVESTIGATE THE EFFICACY OF MANUAL TRACTION ON PAIN AND RANGE OF MOTION IN CERVICAL RADICULOPATHY.
- [Background] Popescu A, Lee H. Neck Pain and Lower Back Pain. Med Clin North Am. 2020 Mar;104(2):279-292. doi: 10.1016/j.mcna.2019.11.003. Epub 2019 Dec 20. PMID 32035569
- [Background] Windsor RE, Malanga G, Benjamin M, Chawla J. Cervical spine anatomy. Medscape; 2017.
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] Sillevis R, Hogg R. Anatomy and clinical relevance of sub occipital soft tissue connections with the dura mater in the upper cervical spine. PeerJ. 2020 Aug 10;8:e9716. doi: 10.7717/peerj.9716. eCollection 2020. PMID 32864219
- [Background] Fredin K, Loras H. Manual therapy, exercise therapy or combined treatment in the management of adult neck pain - A systematic review and meta-analysis. Musculoskelet Sci Pract. 2017 Oct;31:62-71. doi: 10.1016/j.msksp.2017.07.005. Epub 2017 Jul 21. PMID 28750310
- [Background] Rodriguez-Sanz J, Malo-Urries M, Lucha-Lopez MO, Lopez-de-Celis C, Perez-Bellmunt A, Corral-de-Toro J, Hidalgo-Garcia C. Comparison of an exercise program with and without manual therapy for patients with chronic neck pain and upper cervical rotation restriction. Randomized controlled trial. PeerJ. 2021 Nov 24;9:e12546. doi: 10.7717/peerj.12546. eCollection 2021. PMID 34900443
- [Background] Rodriguez-Sanz J, Malo-Urries M, Corral-de-Toro J, Lopez-de-Celis C, Lucha-Lopez MO, Tricas-Moreno JM, Lorente AI, Hidalgo-Garcia C. Does the Addition of Manual Therapy Approach to a Cervical Exercise Program Improve Clinical Outcomes for Patients with Chronic Neck Pain in Short- and Mid-Term? A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Sep 10;17(18):6601. doi: 10.3390/ijerph17186601. PMID 32927858
- [Background] Afzal R, Ghous M, Shakil Ur Rehman S, Masood T. Comparison between Manual Traction, Manual Opening technique and Combination in Patients with cervical radiculopathy: Randomized Control Trial. J Pak Med Assoc. 2019 Sep;69(9):1237-1241. PMID 31511705